CLINICAL TRIAL: NCT01730027
Title: A Randomised, Double Blind, Placebo-Controlled, Multi-Centre, Parallel Group Study to Evaluate the Efficacy and Safety of ADC3680 Administered Once Daily as an Add-On Therapy to Inhaled Corticosteroids and When Co-Administered With Montelukast in Subjects With Inadequately-Controlled Asthma.
Brief Title: A Study to Evaluate Efficacy and Safety of ADC3680 in Subjects With Inadequately-Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmagen Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADC3680-07; 2012-003966-42 (EudraCT Number)
Record Dates: First submitted 2012-11-09; First posted 2012-11-21 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ADC3680 (Experimental): ADC3680 oral once daily
  Interventions: Drug: ADC3680
- Placebo (Placebo Comparator): Placebo oral once daily
  Interventions: Drug: Placebo
- montelukast (Active Comparator): montelukast oral once daily
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: ADC3680 — ADC3680 for 12 weeks plus montelukast for the last 2 weeks of the dosing period
  Arms: ADC3680
Drug: Placebo — Placebo for 12 weeks plus montelukast for the last 2 weeks of the dosing period
  Arms: Placebo
Drug: montelukast — montelukast for 12 weeks
  Arms: montelukast

SUMMARY:
This randomised, double-blind, placebo-controlled study will evaluate the efficacy and safety of ADC3680 administered once daily as an add-on therapy to inhaled corticosteroids and when co-administered with montelukast in patients with inadequately-controlled asthma. Patients will be randomised to 3 Arms to receive ADC3680, placebo or montelukast.

DETAILED DESCRIPTION:
This is a multi-centre, randomised, placebo-controlled, double blind, parallel group 3-arm study (including montelukast as an active comparator) designed to compare the efficacy and safety of a once daily dose of ADC3680 with placebo in subjects with inadequately-controlled asthma despite receiving a low to moderate dose of an ICS controller therapy, over a 10 week treatment period. At the end of the 10 week treatment period open label montelukast (10 mg) will be added to ADC3680 and placebo arms for a two week extension period to assess whether efficacy of ADC3680 is enhanced by the addition of montelukast compared with montelukast alone. The montelukast arm will continue with 10 mg montelukast alone.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years to 50 years (inclusive)
* Diagnosis of asthma (GINA 2011) including a demonstration of reversible airway obstruction
* Pre-bronchodilator FEV1 value ≥ 40% and ≤ 85% of the predicted normal value at baseline
* A score of 1.5 or greater on the Asthma Control Questionnaire at baseline
* Daily use of low to moderate dose of ICS (equivalent to budesonide ≤ 800 µg per day)
* Prescribed a short-acting inhaled bronchodilator as reliever therapy for relief of symptoms
* A peripheral blood eosinophil count ≥ 0.25 x 109/L
* Non-smoker or former smoker who has not smoked in the last six months
* Body mass index (BMI) ≥ 17 and ≤ 35 kg/m2
* Able to comply with the protocol requirements, instructions and restrictions
* Able to provide signed and dated written informed consent

Exclusion Criteria:

* Subjects with severe asthma exacerbation in the 4 weeks prior to consent
* Subjects with respiratory tract infection in the 4 weeks prior to consent
* Subjects with COPD or other relevant lung diseases
* Subjects with clinically significant condition which may compromise subject safety or interfere with study evaluation

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of ADC3680 compared with placebo in improving lung function (FEV1) | 10 weeks
Adding montelukast to ADC3680 in improving lung function (FEV1) | 2 weeks

SECONDARY OUTCOMES:
Efficacy of ADC3680 compared with placebo on mean change in Asthma Control Questionnaire (ACQ) from baseline to Week 10 | 10 weeks
Efficacy of ADC3680 compared with placebo on mean change in trough pre-bronchodilator FEV1 % predicted from baseline to Week 2 | 2 weeks
Efficacy of ADC3680 compared with placebo on mean change in trough pre-bronchodilator FEV1 % predicted from baseline to Week 6 | 6 weeks
Efficacy of ADC3680 compared with placebo on mean change in trough pre-bronchodilator FEV1 % predicted from baseline to Week 10 | 10 weeks
Efficacy of ADC3680 compared with placebo on mean change in post-bronchodilator FEV1 from baseline to Week 10 | 10 weeks
Efficacy of ADC3680 compared with placebo on mean change in pre-bronchodilator PEF (in-clinic) from baseline to Week 2 | 2 weeks
Efficacy of ADC3680 compared with placebo on mean change in pre-bronchodilator PEF (in-clinic) from baseline to Week 6 | 6 weeks
Efficacy of ADC3680 compared with placebo on mean change in pre-bronchodilator PEF (in-clinic) from baseline to Week 10 | 10 weeks
Efficacy of ADC3680 compared with placebo on mean change in blood eosinophils from baseline to Week 10 | 10 weeks
Efficacy of ADC3680 compared with placebo on mean change in serum IgE from baseline to Week 10 | 10 weeks
Adding montelukast to ADC3680 on mean change in ACQ scores from Week 10 to Week 12 | 2 weeks
Adding montelukast to ADC3680 on mean change in trough pre-bronchodilator FEV1 % predicted from Week 10 to Week 12 | 2 weeks
Adding montelukast to ADC3680 on mean change in pre-bronchodilator PEF (in-clinic) from Week 10 to Week 12 | 2 weeks
Adding montelukast to ADC3680 on mean change in blood eosinophils from Week 10 to Week 12 | 2 weeks
Safety of ADC3680 compared to placebo | 10 weeks
  Safety evaluations will include incidence of Serious Adverse Events (from informed consent), severity & frequency of Adverse Events, change in laboratory values (haematology, clinical chemistry and urinalysis), change in vital signs (pulse, systolic and diastolic blood pressure), change in ECG and change in physical examination from baseline to week 10.
Safety of a 2 week administration of ADC3680 in combination with montelukast | 2 weeks
  Safety evaluations will include incidence of Serious Adverse Events, severity & frequency of Adverse Events, change in laboratory values (haematology, clinical chemistry and urinalysis), change in vital signs (pulse, systolic and diastolic blood pressure), change in ECG and change in physical examination from week 10 to week 12.

CONTACTS AND LOCATIONS:
Locations (87):
- United States (35):
  - Pulmagen Investigational Site, Birmingham, Alabama
  - Pulmagen Investigational Site, Huntington Beach, California
  - Pulmagen Investigational Site, Riverside, California
  - Pulmagen Investigational Site, Rolling Hills, California
  - Pulmagen Investigational Site, San Jose, California
  - Pulmagen Investigational Site, Colorado Springs, Colorado
  - Pulmagen Investigational Site, Waterbury, Connecticut
  - Pulmagen Investigational Site, Lawrenceville, Georgia
  - Pulmagen Investigational Site, Eagle, Idaho
  - Pulmagen Investigational Site, Nottingham, Maryland
  - Pulmagen Investigational Site, Plymouth, Minnesota
  - Pulmagen Investigational Site, Bellevue, Nebraska
  - Pulmagen Investigational Site, Brick, New Jersey
  - Pulmagen Investigatinal Site, Clemmons, North Carolina
  - Pulmagen Investigational Site, Canton, Ohio
  - Pulamgen Investigational Site, Cincinnati, Ohio
  - Pulmagen Investigational Site, Maumee, Ohio
  - Pulmagen Investigational Site, Oklahoma City, Oklahoma
  - Pulmagen Investigational Site, Tulsa, Oklahoma
  - Pulmagen Investigational Site, Medford, Oregon
  - Pulmagen Investigational Site, Portland, Oregon
  - Pulmagen Investigational Site, East Providence, Rhode Island
  - Pulmagen Investigational Site, Warwick, Rhode Island
  - Pulmagen Investigational Site, Charleston, South Carolina
  - Pulmagen Investigational Site, Fort Mill, South Carolina
  - Pulmagen Investigational Site, Arlington, Texas
  - Pulmagen Investigational Site, Austin, Texas
  - Pulmagen Investigational Site, Houston, Texas
  - Pulmagen Investigational Site, Killeen, Texas
  - Pulmagen Investigational Site, Waco, Texas
  - Pulmagen Investgational Site, Woodway, Texas
  - Pulmagen Investigational Site, Draper, Utah
  - Pulmagen Investigational Site, Seattle, Washington
  - Pulmagen Investigational Site, Tacoma, Washington
  - Pulmagen Investigational Site, Greenfield, Wisconsin
- Croatia (4):
  - Pulmagen Investigational Site, Čakovec
  - Pulmagen Investigational Site, Sisak
  - Pulmagen Investigational Site, Varaždin
  - Pulmagen Investigational Site, Zagreb
- Czechia (9):
  - Pulmagen Investigational Site, Beroun
  - Pulmagen Investigational Site, Brno
  - Pulmagen Investigational Site, Havlíčkův Brod
  - Pulmagen Investigational Site, Holešov
  - Pulmagen Investigational Site, Jaroměř
  - Pulmagen Investigational Site, Neratovice
  - Pulmagen Investigational Site, Svitavy
  - Pulmagen Investigational Site, Teplice
  - Pulmagen Investigational Site, Třemošná
- Germany (14):
  - Pulmagen Investigational Site, Augsburg
  - Pulmagen Investigational Site, Bad Wörishofen
  - Pulmagen Investigational Site, Berlin
  - Pulmagen Investigational Site, Bonn
  - Pulmagen Investigational Site, Deggingen
  - Pulmagen Investigational Site, Dresden
  - Pulmagen Investigational Site, Geesthacht
  - Pulmagen Investigational Site, Hagen
  - Pulmagen Investigational Site, Hamburg
  - Pulmagen Investigational Site, Hanover
  - Pulmagen Investigational Site, Marburg
  - Pulmagen Investigational Site, Schwerin
  - Pulmagen Investigational Site, Teuchem
  - Pulmagen Investigational Site, Weyhe
- Hungary (7):
  - Pulmagen Investigational Site, Balassagyarmat
  - Pulmagen Investigational Site, Budapest
  - Pulmagen Investigational Site, Kaposvár
  - Pulmagen Investigational Site, Komló
  - Pulmagen Investigational Site, Pécs
  - Pulmagen Investigational Site, Százhalombatta
  - Pulmagen Investigational Site, Szombathely
- Poland (18):
  - Pulmagen Investigational Site, Bialystok
  - Pulmagen Investigational Site, Bielsko-Biala
  - Pulmagen Investigational Site, Bieńkówka
  - Pulmagen Investigational Site, Bydgoszcz
  - Pulmagen Investigational Site, Kielce
  - Pulmagen Investigational Site, Krakow
  - Pulmagen Investigational Site, Lodz
  - Pulmagen Investigational Site, Olsztyn
  - Pulmagen Investigational Site, Ostrow Wilekopolski
  - Pulmagen Investigational Site, Poznan
  - Pulmagen Investigational Site, Proszowice
  - Pulmagen Investigational Site, Skierniewice
  - Pulmagen Investigational Site, Tarnów
  - Pulamgen Investigational Site, Warsaw
  - Pulmagen Investigational Site, Wilkowice-Bystra
  - Pulmagen Investigational Site, Wroclaw
  - Pulmagen Investigational Site, Zabrze
  - Pulmagen Investigational Site, Zgierz